CLINICAL TRIAL: NCT04188977
Title: Facilitating the Implementation of Interim Methadone to Increase Treatment Access: A Multi-Site Implementation Trial
Brief Title: Facilitating the Implementation of Interim Methadone to Increase Treatment Access
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Friends Research Institute, Inc. (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Health Services Research
Other Study IDs: U01DA046910 (NIH); U01DA046910 (NIH)
Record Dates: First submitted 2019-11-12; First posted 2019-12-06 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Opioid-use Disorder
Keywords: Implementation Facilitation; Interim methadone treatment; Opioid Treatment Program
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: Type 3 implementation-effectiveness type study using a modified stepped wedge design
Who Masked: Care Provider
Masking Description: OTPs are masked during their Pre-Implementation Phase.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Practice (Other): OTPs are able to request from state and federal health department officials to utilize interim methadone treatment to address admission delays in their OTP.
  Interventions: Other: Usual Practice
- Implementation Facilitation (Experimental): Implementation Facilitation (IF) will consist of educational outreach to OTP staff, identification of local champions, training, performance feedback, and learning collaborative for OTP staff and state health department officials.
  Interventions: Other: Implementation Facilitation

INTERVENTIONS:
Other: Usual Practice — OTP Directors are able to ask their state health officials permission to use interim methadone treatment. The state officials are in turn able to ask officials from the Center of Substance Abuse Treatment for permission to provide interim methadone treatment.
  Arms: Usual Practice
Other: Implementation Facilitation — Implementation Facilitation (IF) will consist of educational outreach to OTP staff, identification of local champions, training, performance feedback, and learning collaborative for OTP staff and state health department officials.
  Arms: Implementation Facilitation

SUMMARY:
The primary aim of this study is to evaluate the effectiveness of Implementation Facilitation (IF) in promoting increased accessibility to methadone treatment.

DETAILED DESCRIPTION:
This is a Type 3 implementation-effectiveness type study using a modified stepped wedge design. The study's purpose is to examine the effectiveness of Implementation Facilitation (IF) to prompt participating Opioid Treatment Programs (OTPs) to utilize interim methadone treatment and other approaches to reduce OTP admission delays. Interim methadone treamtent is an evidence-based practice permitted under federal OTP regulations to provide methadone treatment without routine counseling for individuals requesting methadone treatment who otherwise would not be able to be admitted to such treatment within 14 days of request. The study will be conducted at six OTPs in the US that are unable to admit individuals within 14 days of their request for methadone treatment. The OTPs will participate in a baseline Pre-Implementation Phase, an Implementation Phase, followed by a Sustainability Phase. OTPs will be randomly assigned in groups of two to the order in which they will initiate the Implementation Phase. IF will be delivered at the level of the OTP staff and their state health department official responsible for OTP oversight. OTP staff and state health department officials will be interviewed regarding facilitators and barriers to implementing interim methadone and other approaches to reduce admission delays. De-identified data will be gathered from the OTPs on the effectiveness of IF in prompting the implementation of interim methadone and reducing admission delays.

ELIGIBILITY:
Inclusion Criteria (Staff):

* OTP staff
* State health department staff responsible for OTP oversight

Exclusion Criteria:

* Unwilling to be interviewed

Inclusion Criteria (OTP applicants):

* requesting admission to OTP

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Accessibility | Nine months
  Accessibility will be assessed from de-identified OTP records as the proportion of individuals requesting methadone treatment who receive at least one dose of methadone through either interim methadone (IM) or standard methadone within 14 days, divided by the number of individuals requesting methadone treatment.

SECONDARY OUTCOMES:
Uptake | Nine months
  Uptake will be assessed from de-identified OTP records as the proportion of individuals unable to gain admission within 14 days who receive at least one interim methadone dose divided by the number of individuals who were unable to be admitted within 14 days.
Efficiency | Nine months
  Efficiency will be assessed from de-identified OTP records as the number of days from the request for OTP admission prior to receiving a first methadone dose.
Fidelity | Six months
  Fidelity will be assessed from de-identified OTP records as the proportion of interim methadone patients transferred to standard methadone treatment within the permitted time limit from starting interim methadone treatment.
Uptake during the Sustainability Phase | Six months
  Sustainability will be assessed from de-identified OTP records as the proportion of interim methadone patients admitted within 14 days of request during the Sustainability Phase
Effectiveness: percentage of opioid positive tests | Six months
  Effectiveness will be assessed from de-identified OTP records as the percentage of opioid-positive urine tests of interim methadone patients at the time of transfer to standard methadone treatment

CONTACTS AND LOCATIONS:
Overall Officials: Robert P Schwartz, M.D., Principal Investigator — Friends Research Institute, Inc.
Locations (1):
- Robert Philip Schwartz, M.D., Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gryczynski J, Mitchell SG, Whitter M, Fuller D, Mitchell MM, Edelman EJ, Schwartz RP. A trial of implementation facilitation to increase timely admission to methadone treatment. J Subst Use Addict Treat. 2024 Jul;162:209375. doi: 10.1016/j.josat.2024.209375. Epub 2024 Apr 19. PMID 38642889
- [Derived] Mitchell SG, Jester J, Gryczynski J, Whitter M, Fuller D, Halsted C, Schwartz RP. Impact of COVID-19-related methadone regulatory flexibilities: views of state opioid treatment authorities and program staff. Addict Sci Clin Pract. 2023 Oct 17;18(1):61. doi: 10.1186/s13722-023-00417-7. PMID 37848970